# W UNIVERSITY of WASHINGTON

# APPLICATION: Continuing Review (Status Report), Renew or Close

Human Subjects Division Box 359470 Seattle, WA 98195-9470 Phone: 206-543-0098

Fax: 206-543-9218

Version 5.1

For instructions on how to complete this form, see the last page.

| For HS | Date Received: | | |
|---|---|---|---|
| [ ] Master Copy | Approved | | RECEIVED Human Subjects Division |
| [ ] IRB Working Copy | [] Disapproved | | |
| [ ] Researcher Copy | [] Withdrawn | | OCT 1 4 2014 |
| [ ] Full IRB Review Required | | | UW |
| Expedited Review | | | DORA CRR # |
| Approval period from: 12-19-14 | | To: 12-18-15 | |
| Date of IRB action: 12-3-1- | | Printed name: Heidi Thielmann | |
| IRB Chair or Designee Signature: | to | | |

| | Research Stud | dy Informat | ion | | |
|---|---|---|---|---|---|
| Submission Reason | [ X] RENEW IRB application | | [ ] CLOSE IRB application | | |
| Expiration date of IRB approval | | | 12/18/2014 | | |
| RB Application # | 43961 | | IRB Committee A | | |
| RB Application Title | Lactobacillus probiotic for | cillus probiotic for prevention of recurrent UTI | | | |
| ead Researcher Name | Ann Stapleton, MD | Contac | Contact Name Position and/or academic appointment | | Niki DeShaw<br>Study Coordinator |
| Position and/or academic appointment | Professor | | | | |
| Department/Division | Med/All & Inf. Diseases | Departm | Department/Division | | Med/All & Inf. Diseases |
| Phone # | 206-616-4121 | Phone # | | 206-685-1048 | |
| ax# | 206-616-4125 | Fax# | | | |
| | 356423 | Campus | Campus Box # | | 354410 |
| Campus Box # Street address, if applicable | 330423 | Street address, if applicable | | | |
| | stapl@uw.edu | Email | The state of the s | | ndeshaw@uw.edu |
| Email | stapi@dw.cdd | Specification | | Fig. 7 | |
| [] Person completing this form is the same as the Lead Researcher | | | on completing thi | s form is t | he same as the Contact |
| Name of Person Completing This Form (If not Lead Researcher or Contact): | | | Email: | | Phone: |
| | Name and Mailing Address for<br>correspondence will be directed to contri | act person, or | r lead researcher | if no conta | act person) |
| Name: | Campus Box#: | Other address if not at U | | V: | |

# A. Research Activity Status

RECEIVED Human Subjects Division

# UNIVERSITY OF WASHINGTON CONSENT FORM

MAR 26 2015

# Lactobacillus Probiotic for Prevention of Recurrent Urinary Tract Infections

Researchers:

Ann Stapleton, MD Professor, Medicine/Infectious Diseases 206-616-4121 Research Study Coord., Medicine/Infectious Dis. 206-685-1048

Ellen Cassen, ARNP Study NP, Medicine/Infectious Diseases 206-685-1048

24-Hour Emergency Contact: 206-598-6190 (UMC operator; ask to have Dr. Stapleton paged)

## Researchers' statement

We are asking you to be in a research study. The purpose of this consent form is to give you the information you will need to help you decide whether to be in the study or not. Please read the form carefully. You may ask questions about the purpose of the research, what we would ask you to do, the possible risks and benefits, your rights as a volunteer, and anything else about the research or this form that is not clear. When we have answered all your questions, you can decide if you want to be in the study or not. This process is called "informed consent." We will give you a copy of this form for your records.

### PURPOSE OF THE STUDY

The purpose of this research is to see whether LACTIN-V (*Lactobacillus crispatus* CTV-05) is an effective method of preventing recurrent urinary tract infections (UTI's) and to learn about the side effects of LACTIN-V. LACTIN-V is a vaginal applicator that contains *Lactobacillus crispatus*, an organism found naturally in the vaginas of healthy women. Lactobacillus bacteria are thought to help prevent other bacteria such as *E. coli* from causing UTI's.

In this study we will compare LACTIN-V with placebo (an inactive vaginal applicator without any medicine). LACTIN-V is an experimental drug. The U.S. Food and Drug Administration (FDA) allow LACTIN-V to be used only in research with a limited number of people. Hall Health Primary Care Center will be the only study site. About 276 people will take part in this study. About 138 participants will receive LACTIN-V and about 138 participants will receive placebo during the study.

#### STUDY PROCEDURES

## Visit 0 (Screening Visit):

If you agree to be in this study, we will ask you to do the following things: First, we will do a screening evaluation. The purpose of the screening evaluation is to find out if you are eligible to be in the study. During this evaluation a study nurse practitioner will ask you some questions about your medical and sexual history and your current symptoms of UTI. Some of the questions are of a personal nature, such as your sexual preference and your total number of

APR 02 2015

lifetime sexual partners. You are free to refuse to answer any question. You will be asked to provide a urine sample to test for infection. A study nurse practitioner will collect vaginal specimens to test for vaginal bacteria and vaginal infections.

The initial study visit will take about one hour. If the results of the screening show that you are eligible for this study, we will ask you to return to the clinic within 3-10 day after completing your UTI treatment for a randomization visit (v1).

## Repository Study:

We will ask you if you want to take part in a separate study for permanent storage of unused samples and study data (including questionnaires, bacteria, and laboratory results) taken as part of this study. We want to save your unused samples and study data to help us understand the reasons why UTIs occur. If you are interested in participation in the repository study, we will go over the "Specimen Repository for UTI Studies" consent form with you. Your participation in the repository study is voluntary. You don't have to give us permission to keep any unused samples and study data as part of the repository study if you don't want us to. We will ask you to mark whether or not you are interested in hearing more about the repository study at the end of the consent form.

## Visit 1 (Randomization Visit):

During this visit, you will be asked about any urinary or vaginal symptoms. You will be asked to provide a urine sample to see if your UTI has resolved and for a pregnancy test. You will be asked to have a physical exam including a pelvic and speculum exam. A study nurse practitioner will collect vaginal specimens to test for vaginal bacteria and vaginal infections.

Next, you will be randomly assigned (like flipping a coin) to use LACTIN-V or placebo vaginal applicators. You will not be told which you will be using, and the researchers will not know until the end of the study. You will not be able to tell which one you are using. Each LACTIN-V applicator contains *Lactobacillus crispatus* CTV-O5 and other preservatives. Each placebo suppository contains other preservatives.

You will be instructed how to use the applicators. You will also be given written instructions on how to use, store, and handle the applicators, and a diary to record when you use the applicators and any symptoms you may have during the study. (You will be given 15 applicators). You will insert 15 applicators during this study. The applicators are to be used daily for five days during the first week and then once per week for 10 weeks starting the second week. To insert an applicator, you will hold one applicator between your thumb and fingers (like a tampon), insert the applicator into the opening of the vagina, and then push the applicator plunger. You will insert the first applicator in the clinic during your visit. You will be asked not to have sexual intercourse or use tampons for 24 hours after inserting an applicator. You will also be asked not to use spermicidal vaginal products. We will also ask you not to take other probiotics (excluding food products) during the study. You will also be asked not to use other vaginal products such as

creams, gels, foams, sponges, lubricants, or douches or take antibiotics for a UTI during this study unless your doctor prescribes it. The visit will take 30-60 minutes.

#### Visits 2-6

We will then ask you to return to the Hall Health clinic in 2 weeks and then once a month for the next 4 months, after your randomization visit. During these visits a study nurse practitioner will ask you about any side-effects you may have had from the study drug or placebo. The study nurse practitioner will also ask you if you have had any UTI's since your last visit. You will be asked to give a urine sample for culture. You will also be asked to have a physical exam, and vaginal tests for infection, lactobacillus (including lactobacillus from LACTIN-V) and *E. coli*. A speculum exam will only be done at your last visit unless you have symptoms of vaginal infection. At the last visit you will have a urine pregnancy test. These visits will take 30 minutes.

### Other Visits:

If you have a UTI or vaginal infection during the study, we will ask you to see us at Hall Health Primary Care Center for treatment. You will be treated with a standard medication at no cost to you. If you have a UTI during the study, you will continue to use the study applicator on schedule.

# RISKS, STRESS, OR DISCOMFORT

As with any drug, there may be side effects, including the risk of death that we do not know about. LACTIN-V is an experimental drug and has only been taken by a limited number of people. Because it is a natural product containing lactobacillus bacteria that are normally found in the vaginas of healthy women, the risk of taking LACTIN-V is expected to be small. Some of the side-effects that might occur include genital and vaginal itching, burning, pain, discharge, odor, vaginal yeast infection, or diarrhea. The risk of rash is expected to be small. The risk of an allergic reaction to LACTIN-V is expected to be small.

Some of the questions you are asked may be sensitive or embarrassing to you. You may refuse to answer any question at any time.

You may experience minor discomfort during pelvic exams, similar to what you would expect from a pelvic exam performed for routine gynecologic care. The urine and vaginal specimen collection should cause minimal discomfort.

We don't know what the effects of LACTIN-V might be on a developing fetus. If you are a woman of childbearing potential, we will test you to make sure you are not pregnant. You must not get pregnant while in this study. You or your sexual partner must use a reliable method of birth control for while you are participating in the study. Reliable methods of birth control include birth control pills, intrauterine device (IUC), implanted contraceptive (such as Norplant),

vasectomy, tubal ligation, Nuva-ring, or condoms (to be provided). Condoms with spermicide cannot be used because spermicide will kill lactobacilli.

If you develop a UTI during the study, you may experience side effects from the antibiotic used for treatment. Common side effects may include nausea, diarrhea, vomiting, abdominal discomfort, rash including sensitivity to sunlight, sleep disturbance, headache, and dizziness. Life-threatening reactions to any antibiotic can rarely occur.

#### ALTERNATIVES TO TAKING PART IN THIS STUDY

There are alternatives to being in this study. For women with frequent UTI's, the alternatives include taking antibiotics to prevent UTI or prompt treatment of UTI's when they reoccur.

#### BENEFITS OF THE STUDY

You may benefit from the study if LACTIN-V proves to be effective. We cannot guarantee that there will be any benefit to you. If you are in the group that takes placebo (inactive substance without medicine), you may experience the risks, stress and discomforts of the interviews, exams, and screening tests, but will not benefit from taking LACTIN-V during the study. We hope that the results of this study will help us find a new safe and effective alternative to antibiotics for the prevention of UTI's in women.

#### MEDICAL RECORD INFORMATION

Policies require that we put information about this research into your permanent medical record at UW Medicine. If you do not have a medical record there, one will be created for you even if your only connection with them is as a research subject.

## Information that will be put into your medical record

1. Your name, address, telephone number, date of birth, social security number, health insurance information, billing information, and any other information you provide on the hospital or clinic information form.

#### Who will have access

This medical record will be permanent. It will be stored with all other UW Medicine medical records. A copy of your record may also be stored on the secure UW Medicine medical record computer system. Access to medical records and the computer system is restricted to only authorized staff with passwords for the system. Only UW Medicine staff and people who have legal access to your medical record will be able to see it. This may include your insurance company and government regulatory agencies. If you have already given permission to anyone (such as your health insurance company) to look at your medical record, they may receive this research information if they ask for a copy of your medical record.

#### SOURCE OF FUNDING

• the federal Food and Drug Administration (FDA), if required by the FDA;

#### OTHER INFORMATION

You may refuse to participate and you are free to withdraw from this study at any time without penalty or loss of benefits to which you are otherwise entitled.

You will not be charged for study related procedures. This includes the research visit, laboratory tests, and antibiotics (if you have symptoms of a UTI)

You will be asked to return all applicators and study diaries. You will be paid \$25 dollars for your screening visit thru visit 5, and \$50 dollars at visit 6 for taking part in this study, as well as returning all study material.

#### COMPENSATION FOR INJURY

If you think you have an injury or illness related to this study, contact Ellen Cassen, ARNP at 206-685-1048 right away. She will treat your or refer you for treatment.

No money has been set aside to pay for things like lost wages, lost time, or pain. However, you do not waive any rights by signing this consent form.

| The UW wi study. | ll pay up to \$10,000 to rein | nburse for treatment of injury or illne | ess resulting from the |
|---|---|---|---|
| Printed Nan | ne of Researcher | Signature of Researcher | Date |
| Subject's Sta | atement | | |
| chance to as<br>researchers the Human S | k questions. If I have questisted above. If I have any of Subjects Division at 206-54 | volunteer to take part in this research tions later about the research, I can a questions about my rights as a resear 3-0098. I give permission to the research form. I will receive a copy of the | sk one of the<br>ch subject, I can call<br>earchers to use my |
| ☐ Yes<br>☐ No | Please indicate whether of the repository study. | not you would be interested hearing | g more about |
| Printed Nam<br>Copies to: | e of Subject<br>Subject | Signature of Subject | Date |

Investigators' file

The study team and the University of Washington are receiving financial support from a National Institutes of Health sponsored grant. The study product is provided by Osel Inc.

#### CONFIDENTIALITY OF RESEARCH INFORMATION

All the information you provide will be confidential. Your name and other identifying information will be linked to a unique study ID. Your study ID will not include any information that can identify you. All of the data we collect from you will be coded with your study ID and kept in a locked cabinet, or password protected computer files. The master list linking your identifying information to your study data will be kept in a separate, secure location. We will destroy the link between your identifying information and study data after the data collection is complete.

The urine samples we collect from you will not include any information that can identify you. They will be coded with your study ID only and stored in a freezer at our UTI research laboratory. Your coded samples will be stored until they are all used up. If you want to withdraw any unused samples from further use, please contact Niki DeShaw at 206-685-1048.

If you give us permission to send your unused samples and study data to other researchers, they will not include any information that can identify you. They will be coded with your study ID only and will be kept indefinitely.

If you agree to take part in the repository study, your study data and samples will be kept indefinitely. More information about the storage of data and samples related to the repository is described in the "Specimen Repository for UTI Studies" consent form.

If we publish the results of this study, we will not use your name or other personal information.

Government or university staff sometimes review studies such as this one to make sure they are being done safely and legally. If a review of this study takes place, your records may be examined. The reviewers will protect your privacy. The study records will not used to put you at legal risk of harm. We have a Certificate of Confidentiality from the federal National Institutes of Health. This helps us protect your privacy. The Certificate means that we do not have to give out identifying information about you even if we are asked to by a court of law. We will use the Certificate to resist any demands for identifying information.

We can't use the Certificate to withhold your research information if you give your written consent to give it to an insurer, employer, or other person. Also, you or a member of your family can share information about yourself or your part in this research if you wish.

There are some limits to this protection. We will voluntarily provide the information to:

- a member of the federal government who needs it in order to audit or evaluate the research;
- individuals at the University of Washington, the funding agency, and other groups involved in the research, if they need the information to make sure the research is being done correctly;